CLINICAL TRIAL: NCT02563782
Title: Ph 2, Double-Masked, Randomized, Parallel, Sham Surgery/Placebo Control, Multi-Center Study to Evaluate Systemic IMT Regimens as Graft Rejection Prophylaxis Following Transplantation of hESC Derived RPE Cells in Patients With AMD
Brief Title: Study to Evaluate Sub-retinal Transplantation of Retinal Pigmented Epithelial Cells in Patients With Dry AMD
Acronym: PORTRAY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Changes to the study design and the cell line
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7317-CL-0002; MA09-hRPE AMD 02 PORTRAY (Other: Sponsor)
Record Dates: First submitted 2015-09-21; First posted 2015-09-30 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Sham Comparator): Sham surgery and placebo immunosuppressive therapy (IMT)
  Interventions: Drug: Placebo tacrolimus and mycophenolate mofetil; Procedure: Sham Surgery
- Active Group (Active Comparator): Sub-retinal transplantation of MA09-hRPE cells and IMT
  Interventions: Biological: Sub-retinal transplantation of MA09-hRPE cells; Drug: tacrolimus and mycophenolate mofetil

INTERVENTIONS:
Biological: Sub-retinal transplantation of MA09-hRPE cells — transplantation
  Arms: Active Group
Drug: tacrolimus and mycophenolate mofetil — Immunosuppressive Agents
  Arms: Active Group
Drug: Placebo tacrolimus and mycophenolate mofetil — placebo
  Arms: Control group
Procedure: Sham Surgery — Sham surgery
  Arms: Control group

SUMMARY:
To evaluate the safety of 3 regimens of short-term, low-dose systemic IMT as rejection prophylaxis prior to and/or following transplant of MA09-hRPE cells.

DETAILED DESCRIPTION:
This study will be a Phase 2, double-masked, randomized, parallel group, sham surgery/placebo control, multi-center trial. Subjects will be randomized in a 3:1 ratio to either the treatment or control group respectively. Subjects randomized to the treatment group will receive transplantation with 200,000 MA09-hRPE (human embryonic stem cell derived retinal pigmented epithelial)cells in one eye. Subjects randomized to the control group will have a sham surgery without transplantation of MA09-hRPE cells. The study eye must meet all eligibility criteria. If both eyes meet all eligibility criteria, then the study eye will be the eye with the worst Best Corrected Visual Acuity (BCVA) score at screening. If both eyes have identical BCVA scores, then the study eye will be chosen by the Investigator and the subject. There will be 3 cohorts, each with a different regimen of low-dose IMT [tacrolimus and mycophenolate mofetil (MMF)]. Subjects will be randomized to treatment or control within cohorts, defined by severity of BCVA in the study eye at Screening. Enrollment in Cohort 1 and 2 will be concurrent. Enrollment into Cohort 3 will begin once Cohort 2 is fully enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Geographic atrophy (GA) secondary to AMD with no evidence of prior to active choroidal neovascularization (CNV) in the study eye.
* BCVA in the study eye must be between 4 and 58 Early Treatment of Diabetic Retinopathy Study (EDTRS) letters (20/800 to 20/80; 0.025-0.25)
* Subjects must be willing to take IMT and willing to discontinue any medication that has a known strong interaction with tacrolimus or mycophenolate mofetil (MMF)

Exclusion Criteria:

* Macular atrophy due to causes other than AMD
* Other sight-threatening ocular disease
* Current or prior history of optic neuropathy, retinal dystrophy, retinitis pigmentosa, chorioretinitis, vasoocclusive disease, retinal vascular disease or retinal degenerative disease OTHER than AMD
* History of uveitis
* History of allergic reaction to sulfa drugs
* Solid organ or bone marrow transplant recipient
* History of malignancy within the previous 5 years (except for BCC (basal cell carcinoma), SCC (squamous cell carcinoma) or in-situ cervical)
* History of myocardial infarction with past 12 months
* History of clinically significant cardiac dysrhythmia
* History of diabetes mellitus, bowel disease, tuberculosis
* Prior treatment for non-exudative AMD
* Intraocular, refractive or cataract surgery in the last 12 weeks
* Prior retinal surgery, vitrectomy, macular laser photocoagulation, external beam radiation therapy, transpupillary thermotherapy, glaucoma filtration surgery or corneal surgery (except cataract surgery)
* Receipt of gene transfer of cell transplant therapy in a prior clinical trial
* Participation in any other interventional clinical trial within the last 12 weeks

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with evidence of graft failure or rejection. | 18 months

SECONDARY OUTCOMES:
Change in area of geographic atrophy by Optical coherence tomography | 18 months
  Change from baseline to Week 78
Change in area of geographic atrophy by Autofluorescence | 18 months
  Change from baseline to Week 78
Change in average Best Corrected Visual Acuity (BCVA) | 18 months
  Change from baseline to Week 78

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided